CLINICAL TRIAL: NCT04729023
Title: The Effect of Pars Plana Vitrectomy Combined With Phacoemulsification Cataract Surgery in Phakic Diabetes Retinopathy Patients Over 45 Years Old: a Multicenter Randomized Controlled Clinical Study
Brief Title: Pars Plana Vitrectomy Combined With Phacoemulsification Cataract Surgery in Phakic Diabetes Retinopathy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020KYPJ167
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Diabetic Retinopathy; Diabetic Cataract
Keywords: Diabetic Retinopathy; Diabetic Cataract; Pars plana vitrectomy; Phacoemulsification
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined surgery group (Experimental): In this group, all eligible patients will receive pars plana vitrectomy combined with phacoemulsification cataract surgery.
  Interventions: Procedure: Pars plana vitrectomy combined with cataract surgery.
- Subsequent surgery group (Active Comparator): In this group, all eligible patients will receive pars plana vitrectomy first. And a subsequent phacoemulsification will be systematically performed 6 months after the PPV surgery.
  Interventions: Procedure: Pars plana vitrectomy with subsequent cataract surgery.

INTERVENTIONS:
Procedure: Pars plana vitrectomy combined with cataract surgery. — In the combined surgery group, phakic diabetes retinopathy patients over 45 years old without severe lens opacity will receive pars plana vitrectomy combined with phacoemulsification and intraocular lens (IOL) implantation at the same time.
  Arms: Combined surgery group
Procedure: Pars plana vitrectomy with subsequent cataract surgery. — In the control group, phakic diabetes retinopathy patients over 45 years old without severe lens opacity will first receive pars plana vitrectomy and a subsequent phacoemulsification with IOL implantation will be performed at least 6 month after the PPV.
  Arms: Subsequent surgery group

SUMMARY:
Pars plana vitrectomy (PPV) is one of the most widely used surgical therapies to proliferative diabetic retinopathy in the world.

However, as a predictable consequence of PPV surgery, postoperative cataract is observed in 79%-95% of phakic diabetes retinopathy patients after PPV in 6-24 months and a subsequent cataract surgery is usually required. While, the subsequent cataract surgeries not only bring additional economy and workload burden, but also increase the surgical risks. Since the two-step surgical approach has its defects, the combination of PPV and phacoemulsification is an ideal surgical option.

This study is a multi-center prospective study, aimed to evaluate the effect of PPV combined with phacoemulsification cataract surgery in phakic diabetes retinopathy patients, and make a comparation between the combined surgery and the two-step surgery in patients without severe lens opacities.

DETAILED DESCRIPTION:
The prevalence of diabetes retinopathy is increasing dramatically recent years. Pars plana vitrectomy (PPV) is one of the most widely used surgical therapies to proliferative diabetic retinopathy in the world.

However, as a predictable consequence of PPV surgery, postoperative cataract is observed in 79%-95% of phakic diabetes retinopathy patients after PPV in 6-24 months.Generally, subsequent cataract surgeries are required for the phakic patients within 6-16 months after the PPV surgery to improve visualization. While, the subsequent cataract surgeries not only bring additional economy and workload burden, but also increase the surgical risks because of the deep anterior chamber, zonular dehiscence, and inflammation. Since the two-step surgical approach has its defects, the combination of PPV and phacoemulsification is an ideal surgical option, which is only suggested in patients with severe lens opacities before the PPV surgery so far. For those with mild-moderate lens opacities, the benefits of combined surgery is unknown.

This study is a multi-center prospective study, aimed to evaluate the effect of PPV combined with phacoemulsification cataract surgery in phakic diabetes retinopathy patients, and make a comparation between the combined surgery and the two-step surgery in patients without severe lens opacities.

ELIGIBILITY:
Inclusion Criteria:

1. Proliferative diabetes retinopathy ;
2. Age over 45 years old;
3. mild-moderate lens opacities(LOCSⅢ : C3N3P3 or below);
4. recognition of at least one alphabet in ETDRS chart.

Exclusion Criteria:

1. Long-standing retinal detachment (more than three months), macular affected
2. Low Vision or blind on the other eye;
3. Macular degeneration, including age-related macular degeneration and Polypoidal choroidal vasculopathy;
4. Ocular trauma;
5. Glaucoma;
6. Hereditary retinopathy;
7. Severe lens opacities before the surgery (LOCSⅢ : C4N4P4 or above).

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Best correct visual acuity (BCVA) | Change from Baseline at 1 week after the surgery(s)
  BCVA with early treatment diabetic retinopathy study (ETDRS) letters
Best correct visual acuity | Change from Baseline at 1 month after the surgery(s)
  BCVA with ETDRS letters
Best correct visual acuity | Change from Baseline at 3 months after the surgery(s)
  BCVA with ETDRS letters
Best correct visual acuity | Change from Baseline at 6 months after the surgery(s)
  BCVA with ETDRS letters

SECONDARY OUTCOMES:
VFQ-25 score | Change from Baseline at 6 months after the surgery(s).
  Visual Function Questionnaire-25, values from 0-100, the higher scores mean a better outcome
Complications | through study completion, an average of 1 year
  Common complications after the surgery like glaucoma, macular edema, iritis, et. al.
Treatment costs | through study completion, an average of 1 year
  The amount of money paid on the surgery(s) by each patient.
Working delay time | through study completion, an average of 1 year
  The working delay time due to the surgery(s).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novak MA, Rice TA, Michels RG, Auer C. The crystalline lens after vitrectomy for diabetic retinopathy. Ophthalmology. 1984 Dec;91(12):1480-4. doi: 10.1016/s0161-6420(84)34100-8. PMID 6521988
- [Background] Hsuan JD, Brown NA, Bron AJ, Patel CK, Rosen PH. Posterior subcapsular and nuclear cataract after vitrectomy. J Cataract Refract Surg. 2001 Mar;27(3):437-44. doi: 10.1016/s0886-3350(00)00585-x. PMID 11255058
- [Background] Melberg NS, Thomas MA. Nuclear sclerotic cataract after vitrectomy in patients younger than 50 years of age. Ophthalmology. 1995 Oct;102(10):1466-71. doi: 10.1016/s0161-6420(95)30844-5. PMID 9097793
- [Background] Blodi BA, Paluska SA. Cataract after vitrectomy in young patients. Ophthalmology. 1997 Jul;104(7):1092-5. doi: 10.1016/s0161-6420(97)30180-8. PMID 9224458
- [Background] Westesson PL, Lundh H. Temporomandibular joint disk displacement: arthrographic and tomographic follow-up after 6 months' treatment with disk-repositioning onlays. Oral Surg Oral Med Oral Pathol. 1988 Sep;66(3):271-8. doi: 10.1016/0030-4220(88)90230-7. PMID 3174063
- [Background] Soto-Hernandez JL, Nunley D, Gutierrez CC, Berk SL. Listeria monocytogenes peritonitis. Am J Gastroenterol. 1988 Feb;83(2):180-2. PMID 3341344
- [Background] Peyman GA, Huamonte F, Goldberg MF. Management of cataract in patients undergoing vitrectomy. Am J Ophthalmol. 1975 Jul;80(1):30-6. doi: 10.1016/0002-9394(75)90864-8. PMID 1155546
- [Background] Treumer F, Bunse A, Rudolf M, Roider J. Pars plana vitrectomy, phacoemulsification and intraocular lens implantation. Comparison of clinical complications in a combined versus two-step surgical approach. Graefes Arch Clin Exp Ophthalmol. 2006 Jul;244(7):808-15. doi: 10.1007/s00417-005-0146-9. Epub 2005 Dec 3. PMID 16328429
- [Background] Biro Z, Kovacs B. Results of cataract surgery in previously vitrectomized eyes. J Cataract Refract Surg. 2002 Jun;28(6):1003-6. doi: 10.1016/s0886-3350(02)01237-3. PMID 12036644
- [Background] Meyers SM, Klein R, Chandra S, Myers FL. Unplanned extracapsular cataract extraction in postvitrectomy eyes. Am J Ophthalmol. 1978 Nov;86(5):624-6. doi: 10.1016/0002-9394(78)90179-4. PMID 309730
- [Background] Smiddy WE, Stark WJ, Michels RG, Maumenee AE, Terry AC, Glaser BM. Cataract extraction after vitrectomy. Ophthalmology. 1987 May;94(5):483-7. doi: 10.1016/s0161-6420(87)33420-7. PMID 3601363
- [Background] Senn P, Schipper I, Perren B. Combined pars plana vitrectomy, phacoemulsification, and intraocular lens implantation in the capsular bag: a comparison to vitrectomy and subsequent cataract surgery as a two-step procedure. Ophthalmic Surg Lasers. 1995 Sep-Oct;26(5):420-8. PMID 8963856
- [Background] Silva PS, Diala PA, Hamam RN, Arrigg PG, Shah ST, Murtha TL, Schlossman DK, Cavallerano JD, Sun JK, Aiello LP. Visual outcomes from pars plana vitrectomy versus combined pars plana vitrectomy, phacoemulsification, and intraocular lens implantation in patients with diabetes. Retina. 2014 Oct;34(10):1960-8. doi: 10.1097/IAE.0000000000000171. PMID 24830822